CLINICAL TRIAL: NCT07288294
Title: Primary-Care Strategies to Enhance Weight Management (PRISM) After Discontinuation of Anti-Obesity Medications
Brief Title: PRImary Care Strategies for Weight Management (PRISM) Study
Acronym: PRISM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORA#24011905
Record Dates: First submitted 2025-11-14; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This project is a randomized feasibility study with a run-in period
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRISM Program (Experimental)
  Interventions: Behavioral: PRISM Program
- Usual Care (No Intervention): Participants will continue to receive their regular, usual primary care.

INTERVENTIONS:
Behavioral: PRISM Program — This is a novel, remotely delivered, self-tailored intervention for post-anti-obesity medication discontinuation weight management. The program incorporates standard-of-care behavioral intervention strategies for weight control to improve routine self-weighing, dietary self-monitoring, and increasing physical activity. The program includes an enhanced focus on strategies to reduce food cue reactivity. The program includes six monthly one-on-one sessions between study staff and participants, asynchronous online check-ins weekly for 12 weeks, and bi-weekly for 12 weeks.
  Arms: PRISM Program

SUMMARY:
The goal of this clinical trial pilot is to determine the feasibility of an intervention to enhance weight management in patients who have stopped taking anti-obesity/weight management medications in primary care. The main questions it aims to answer are:

* Can patients be recruited into the study efficiently?
* Is the program acceptable to patients?
* Can the study be conducted efficiently?

The new program will be compared to usual care.

Participants will be asked to 1) complete short surveys about their medication use while taking the weight management medication, 2) complete online visits using study-provided scales, and 3) complete video visits with study staff monthly and online check-ins weekly, if assigned to the active treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Obesity (body mass index ≥30 kg/m2 or ≥27 kg/m2 with obesity-related comorbidity or self-identified Asian race)
2. For run-in: prescribed liraglutide, semaglutide, or tirzepatide or newer medication approved by the FDA for long-term use for obesity treatment by a primary care provider at Rush University System for Health and have received at least one dose of the medication concurrent with enrollment in the study.
3. For randomization: discontinue their prescribed anti-obesity medication.
4. Age 18+

Exclusion Criteria:

1. Not fluent in English
2. Diagnosis of diabetes (type 1 or type 2)
3. Current or planned pregnancy
4. Bariatric surgery in the past 2 years or planned bariatric surgery.
5. Body mass index ≥60 kg/m2, due to increased injury risk with exercise
6. Body weight ≥ 375 pounds (scale capacity with a margin for regain)
7. No access to home WIFI or a smartphone with data available
8. Medical contraindications to treatment, including significant cognitive impairment, active substance abuse based on the World Health Organization's ASSIST screener, or serious medical illness (e.g., stage 3 or 4 heart failure, cancer, renal failure, etc.)
9. Concurrent engagement with other behavioral treatments for obesity (for randomized phase only).
10. Medication obtained from online/compound pharmacies or prescription from specialty clinic without a prescription from primary care team at the time of enrollment
11. Another member of the household is enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  The recruitment rate will be defined as the number of participants randomized into the clinical trial per month.
Acceptability of the Intervention | 3 and 6 months post randomization
  Self-reported Likert scale items will assess the overall satisfaction with the program, the likelihood participants would recommend the program to others, and their satisfaction with individual treatment components (e.g., the online check-ins).

SECONDARY OUTCOMES:
Medication adherence duration questions | From consent to reported discontinuation, up to 22 months
  A published measure will be used to assess adherence throughout the run-in period. These questions will be asked bi-weekly to assess adherence with minimal participant burden.
Reasons for Discontinuation questions | Baseline
  A published measure will be used to assess reasons for discontinuation throughout the run-in period. These items will be asked only if participants indicate nonadherence.

OTHER OUTCOMES:
Recruitment efficiency | Baseline
  Recruitment efficiency will be defined as the days between the participant's last AOM dose and the date of randomization into the trial.
Retention to the study | 6 months post-randomization
  Retention to the study will be defined as an observed weight assessed during the 6-month assessment period.
Intervention adherence | Randomization to 6 months
  Intervention adherence will be defined as the number of one-on-one intervention sessions completed (out of 6 possible) and the number of online check-ins completed (out of 16).
Percent weight change | 3 and 6 months post-randomization
  Weight data for outcome assessments (0, 3, and 6 months) will be collected remotely.
Adherence to dietary self-monitoring | Randomization to 6 months
  Active treatment arm only: portion of days adherent to self-monitoring recommendations
Physical activity | Randomization to 6 months
  Active treatment arm only: wearable tracking device will monitor their steps per day and minutes of medium and high-intensity activity as determined by the Fitbit algorithm.
Self-weighing frequency | Randomization to 6 months
  A smart scale will be used to collect the frequency of self-weighing behavior. Participants will consent to the electronic scale being used to monitor their weighing behavior. Staff will monitor the days per week of recorded weights and the value of the weights to examine weighing and weight trends.
Intervention staff time | Randomization to 6 months
  Staff will track the time spent conducting and scheduling intervention contacts, including time related to the one-on-one sessions and any additional support provided to participants.
Trial protocol staff time | Baseline to 6 months
  Staff will track their time conducting recruitment efforts, consent visits, and conducting and scheduling assessment appointments.

IPD SHARING:
Plan to Share IPD: Yes